CLINICAL TRIAL: NCT00189657
Title: 5FU/VL Vs LV5FU2 + CPT11 in Stage II-III Resected Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Européenne de Recherche en Oncologie (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AERO-R98
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-09

CONDITIONS: Cancer of the Rectum
MeSH Terms: conditions — Rectal Neoplasms | interventions — Irinotecan

INTERVENTIONS:
Procedure: 5FU/LV Mayo Clinic or LV5FU2
Procedure: LV5FU2 + irinotecan

SUMMARY:
The main objective of this randomized trial is to compare 5FU/LV (Mayo-Clinic regimen or LV5FU2) to LV5FU2 + irinotécan in patients with resected B2 and C rectal cancer. Preoperative radiotherapy is recommended but not mandatory. Main endpoint is disease free survival. Secondary endpoint are overall survival, time to local recurrence, time to distant metastases, and tolerance. A total of 600 patients will be included in the trial.

ELIGIBILITY:
Inclusion Criteria:

* rectal adenocarcinoma
* R0 surgery
* T3, N0, M0 or T4, N0, M0 or N1,2, M0
* chemotherapy can be started within 8 weeks after surgery
* Age > 18
* Performance status ECOG < 3
* preoperative radiotherapy allowed
* preoperative chemotherapy with 5FU +/- LV allowed
* Neutrophiles > 1 500/mm3; Pl. > 100 000/mm3
* Transaminases < 2 x UNL; Alcalines Phosphatases < 2 x UNL; Bili < 1.1 UNL
* creatininemia < 120 µmol/l and/or clearance of creatininemia > 60 ml/mn
* Written informed consent before inclusion

Exclusion Criteria:

* postoperative radiotherapy
* Distant metastases
* Contraindication to any drug contained in the chemotherapy regimens
* Any serious active disease or co-morbid medical condition including digestive inflammatory disease
* Gilbert disease
* severe toxicity of radiotherapy
* Pregnancy or breast feeding
* Absence of contraception in non menopausal women
* Adult patient unable to give informed consent because of intellectual impairment
* Concomitant participation to another trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Piedbois, MD, Principal Investigator — Association Europeenne de Recherche en Oncologie; Thierry Andre, MD, Principal Investigator — GERCOR - Multidisciplinary Oncology Cooperative Group; Alain Piolot, MD, Principal Investigator — Association Europeenne de Recherche en Oncologie; Emmanuel Achille, MD, Principal Investigator — GERCOR - Multidisciplinary Oncology Cooperative Group; Iradj Bobhani, MD, Principal Investigator — Fondation Française de Cancérologie Digestive; Jean-Yves Douillard, MD, Principal Investigator — UNICANCER
Locations (1):
- AERO, Créteil, France